CLINICAL TRIAL: NCT02237430
Title: Randomized Comparison of MynxGrip Vascular Closure Device and Manual Compression for Closure After Femoral Access Angiography. The Closure Devices Used in Every Day Practice Study, CLOSE-UP III Trial
Acronym: CLOSE-UP III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital Skejby (Other)
Collaborators: Vingmed Danmark A/S (Individual)
Responsible Party: Principal Investigator, Evald Hoej Christiansen, MD, Aarhus University Hospital Skejby
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLOSE-UP III
Record Dates: First submitted 2014-09-04; First posted 2014-09-11 (Estimated); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Coronary Disease
Keywords: Coronary angiography (CAG)
MeSH Terms: conditions — Coronary Disease | interventions — Vascular Closure Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Manuel compression (Active Comparator): Conventional manual compression
  Interventions: Other: Manual compression
- MynxGrip closure device (Experimental): Closure device for femoral artery access closure
  Interventions: Device: MynxGrip

INTERVENTIONS:
Device: MynxGrip — Closure device for femoral artery access closure
  Other Names: Closure device
  Arms: MynxGrip closure device
Other: Manual compression — Conventional manual compression
  Arms: Manuel compression

SUMMARY:
Is the MynxGrip (test device) non-inferior to manuel compression (standard comparator) in the incidence of adverse access site related events in-hospital, at 30 days and at 6 months.

DETAILED DESCRIPTION:
Prospective, randomized (1:1), controlled, non-blinded, single center study in 2000 patients comparing the MynxGrip (test device) and manuel compression (standard comparator). Safety and efficacy endpoints will be reported for in-hospital, 30 days and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* >18 year
* Should be able to provide valid informed signed consent
* CAG, possibly including intracoronary measurement (FFR) or intracoronary imaging (IVUS, optical coherence tomography (OCT), NIRS)

Exclusion Criteria:

* Percutaneous coronary intervention (PCI) procedure and/or implantation of stents
* ST-Elevations Myocardial Infarction (STEMI)
* Multiple punctures
* Active infection
* Groin haematoma before the closure procedure
* Known pseudoaneurysm or arteriovenous (AV) fistula in the ipsilateral groin
* Cardiogenic shock
* Prior peripheral arterial surgery in abdomen or lower extremities
* Sheat size >7 F
* Life expectancy less than one year
* Possible pregnancy or positive pregnancy test or breastfeeding women
* Simultaneous or planned subsequent femoral vein access
* Allergy to any of the components in the closure material left in the groin
* Puncture or closure with closure device at same site < 30 days
* Puncture or closure with manuel compression at same site < 5 days
* Patients with peripheral artery disease can be included at operators discretion except if heavy calcification is present at the access site, which at the operators discretion precludes insertion of the closure device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 869 (Actual)
Dates: Start 2014-06-16 (Actual); Primary Completion 2017-05-16 (Actual); Study Completion 2018-12-16 (Actual)

PRIMARY OUTCOMES:
Incidence at 30 days of the composite endpoint of serious access site related major adverse vascular events (MAVE) | 30 days
  This includes: Major bleeding and/or blood transfusion, pseudoaneurysm with indication for treatment, arteriovenous fistula, groin surgery of leg, definitely or possible can be related to the closure procedure, infection needing antibiotics.

SECONDARY OUTCOMES:
Time (min) to haemostasis | 30 days
  From inserting the device (MynxGrip) until haemostasis and from beginning of manual compression to immediately haemostasis
Device failure | 30 minutes
Vasovagal reaction until 5 minutes after end of closure procedure | 30 minutes
Need for new onset of manual compression | 30 days
Pain and discomfort related to the closure procedure | Closure procedure and 30 days
  Assessed on a numerical rating scale (NRS) from 0 (no pain or discomfort) to 10 (worst possible pain or discomfort).
Time to mobilization | participants will be followed for the duration of hospital stay, an expected average of 2 days
  From start of closure procedure to patient is mobilised.
In-hospital large groin haematoma | Participants will be followed for the duration of hospital stay, an expected average of 2 days
  Larger than 5 x 5 cm measured by ruler in the catheterisation laboratory or at discharge
Bleedings according to the Bleeding Academic Research Consortium (BARC) definitions | 1 hour and 30 days
Major bleeding and/or bleeding necessitation blood transfusion | 30 days and 6 months
Pseudoaneurysm with indication for treatment | 30 days and 6 months
Arteriovenous fistula | 30 days and 6 months
Groin surgery and/or possible related vascular surgery | 30 days and 6 months
Infection needing antibiotics | 30 days and 6 months
Need for medical evaluation of possible closure procedure related symptom(s) | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Evald H Christiansen, MD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus N, Denmark

REFERENCES:
- [Derived] Jakobsen L, Holm NR, Maeng M, Thim T, Kristensen SD, Mogensen LH, Christiansen EH. Comparison of MynxGrip vascular closure device and manual compression for closure after femoral access angiography: a randomized controlled trial: the closure devices used in every day practice study, CLOSE-UP III trial. BMC Cardiovasc Disord. 2022 Feb 23;22(1):68. doi: 10.1186/s12872-022-02512-0. PMID 35196986